CLINICAL TRIAL: NCT04001088
Title: The Effects of a Novel Probiotic Supplement on Menopausal Symptoms and Bone Health: A Randomized, Double-blind, Parallel, Placebo-Controlled, Multi-Centre Study
Brief Title: The Effects of a Novel Probiotic Supplement on Menopausal Symptoms and Bone Health
Acronym: MPS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lallemand Health Solutions (Industry)
Collaborators: Nutrasource Pharmaceutical and Nutraceutical Services, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MPS
Record Dates: First submitted 2019-06-25; First posted 2019-06-27 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: Menopause
Keywords: Probiotics; Menopausal symptoms; Bone health; Vulvar and vaginal atrophy; Vaginal microflora; Anxiety; Depression; Urinary incontinence; Metabolic syndrome biomarkers; Sleep quality; Gut microflora; Bone resorption markers; Bone formation markers; Bone Mineral Density (BMD); Fracture risk assessment
MeSH Terms: conditions — Anxiety Disorders; Depression; Urinary Incontinence; Sleep Initiation and Maintenance Disorders | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Probiotics in a capsule.
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Non active ingredients in a capsule.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Dosing regimen of one capsule daily for a maximum of 48 weeks.
  Arms: Probiotic
Other: Placebo — Dosing regimen of one capsule daily for a maximum of 48 weeks.
  Arms: Placebo

SUMMARY:
This Phase II study is designed to evaluate the potential effects of a novel probiotic supplement on the severity of global menopause symptoms (e.g., psychological, somatic, urogenital symptoms) and on bone health in postmenopausal women.

DETAILED DESCRIPTION:
Menopause is a natural phase in which a woman's menstrual cycle permanently cease. During this time, women undergo many biological changes, including a decline of estrogen level or alterations in the vaginal microflora. This can result in the onset of various physiological and psychological menopause-related symptoms which may continue into postmenopausal years.

The present study aims to evaluate the potential effects of a probiotic supplement on global menopause symptoms including psychological, somatic and urogenital symptoms. It is hypothesized that this probiotic, consumed over a 12-week period, will help reduce the symptoms of menopause by modulating the mucosal microflora of the vaginal linings. Additionally, it is hypothesized that the continued consumption of this probiotic combination over a total of 48 weeks will aid in the overall maintenance of bone health and may ameliorate bone density loss.

144 healthy postmenopausal women (≥ 40 to < 60 years old) in the U.S. who are experiencing menopause-related symptoms will be randomized to the study (12-week period), and a subset (72 postmenopausal women) will continue the study for an additional 36 weeks (Bone Health Study).

ELIGIBILITY:
Inclusion Criteria:

* Healthy post-menopausal woman
* Last menstrual period has occurred at least 12 months prior to screening
* ≥40 to <60 years old
* Vaginal pH ≥ 5
* MRS score ≥ 20
* Willing and able to give written informed consent
* Willing to consume IP or placebo, complete questionnaires, records, and daily diaries associated with the study and to complete all clinical study visits
* Willingness to discontinue consumption of probiotic supplements and food containing added probiotics and/or prebiotics (e.g. yogurts with live, active cultures or supplements) o Note: Screened participants will be eligible to participate after completing a 4-week wash-out period.

Exclusion Criteria:

* Milk or soy allergy
* Women with induced menopause through full or partial hysterectomy, chemotherapy or radiation
* Consumption of natural health products used to treat menopausal symptoms such as phytoestrogens, Black Cohosh, dehydroepiandrosterone (DHEA), Dong Quai, vitamin E (>250 IU/day), high consumption of soy food products, unless a 1-month wash-out period has been completed prior to study commencement
* Currently undergoing or have previously undergone HT for treatment of menopausal symptoms, unless a three-month washout has been completed prior to study commencement
* Active vaginal infections/abnormalities (e.g. active urinary tract infection (UTI), genital hemorrhage of unknown origin)

  o Note: Screened participants with infections would be eligible to participate 4 weeks after completing their course of treatment (wash-out period).
* Use of any vaginal medication, vaginal rinses and/or moisturizers, gels containing xylocaine or other analgesic products to decrease pain during intercourse, 1 week before and during study
* Use of any antibiotic drug within 1 month of screening

  o Note: Screened participants could be eligible to participate after a 2-week wash-out period.
* Participants previously diagnosed with hyperparathyroidism and/or hyperthyroidism
* Participation in other clinical studies in the past 6 months
* History of alcohol or drug abuse in the 12 months prior to screening
* History of cancer (except localized skin cancer without metastases) within five (5) years prior to screening
* History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the potential subject at risk because of participation in the study, or influences the results or the potential subject's ability to participate in the study
* History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs (i.e. Crohn's disease, short bowel, acute or chronic pancreatitis or pancreatic insufficiency)
* History of a surgical procedure for the treatment of obesity (e.g., gastric bypass, gastric banding)
* Currently consuming more than 2 standard alcoholic beverages a day. A standard alcoholic beverage is defined as 12 ounces of beer, five (5) ounces of wine, or 1.5 ounces of liquor
* Difficulty swallowing large pills or large quantities of pills
* Any condition or abnormality that, in the opinion of the investigator, would compromise the safety of the subject or the quality of the study data

Ages: 40 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2020-11-18 (Actual); Study Completion 2021-04-23 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the global Menopause Rating Scale (MRS) score | Measured on weeks -2 (screening visit), 0, 4, 8, 12, and 48.
  Assessed using Menopause Rating Scale (MRS) rating scale. 11 questions on a scale from no complaints (0) to very severe symptoms (4). Subscores are added to create a composite or total score. A higher score indicates a greater severity of menopausal symptoms.

SECONDARY OUTCOMES:
Change from baseline in individual components of the Menopause Rating Scale (MRS) (psychological, somatic and urogenital symptoms) | Measured on weeks -2 (screening visit), 0, 4, 8, 12, and 48.
  Assessed using Menopause Rating Scale (MRS) rating scale. 11 questions on a scale from no complaints (0) to very severe symptoms (4). Subscores are added to create the 3 dimensions scores. A higher score indiactes a greater severity of perceived menopausal symptoms.
Change from baseline in vaginal pH | Measured on weeks -2 (screening visit), 0, and 12.
  Vaginal swabs will be collected for pH testing, using pH strips for screening and to measure evolution of pH throughout first part of the study.
Change from baseline in vaginal microbiota | Measured on weeks 0 and 12.
  Effects of the probiotic intervention on overall microbiota composition will be assessed with a vaginal swab. In addition, recovery of the probiotic strains in the vaginal samples will be assessed.
Change from baseline in the Patient Health Questionnaire (PHQ-9) total score | Measured on weeks 0, 4, 8, 12, and 48.
  Depression measured with the Patient Health Questionnaire (PHQ-9). 10 questions. The first 9 questions are on a scale from not at all bothered by symptoms (0) to bothered by symptoms nearly everyday (3). To arrive at the total score, the individual question scores are added. A score of 5-9 indicates minimal symptoms, a score of 10-14 indicates minor depression, dysthymia, or mild Major Depression, a score of 15-19 indicates moderately sever Major Depression and a score of greater than 20 indicates severe Major Depression.
Change from baseline in the Pittsburgh Sleep Quality Index (PSQI) global score | Measured on weeks 0, 4, 8, 12, and 48.
  Sleep quality measured by the Pittsburgh Sleep Quality Index (PSQI). 9 questions. It consists of seven components including: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medications, and daytime dysfunction. Each component score ranges from 0 to 3, whereby 3 reflects the negative extreme, for a global score range of 0 to 21. A score of 5 or greater indicates the reporter has poor sleep quality.
Change from baseline in the Vulvovaginal Symptoms Questionnaire (VSQ) total score. | Measured on weeks 0, 4, 8, 12, and 48.
  Vulvar and vaginal atrophy measured with the Vulvovaginal Symptoms Questionnaire (VSQ). 21 yes (1) or no (0) questions in 4 scales: Symptoms, Emotions, Life-impact, Sexual impact. Total score will be the sum of the first 17 questions if non-sexually active or of the 21 questions if sexually active. A higher score indicates a greater severity of vulvar and vaginal atrophy.
Change in baseline in the Michigan Incontinence Symptom Index (M-ISI) mean score | Measured on weeks 0, 4, 8, 12, and 48.
  Urinary incontinence measured with the Michigan Incontinence Symptom Index (M-ISI). 10 questions with different scales all numbered 0-4. The total score is derived from taking the mean of the 10 reported scores. A higher score indicates a higher severity of incontinence.
Change from baseline in the Generalized Anxiety Disorder-7 (GAD-7) total score | Measured on weeks 0, 4, 8, 12, and 48.
  Anxiety measured with the Generalized Anxiety Disorder-7 (GAD-7). 7 questions scaled from not at all sure (0) to nearly every day (3). Total score is derived from the addition of answer to each question. A higher score indicates a higher level of detected anxiety.

OTHER OUTCOMES:
Change from baseline in levels of Metabolic Syndrome biomarkers (serum cholesterol [total, LDL, HDL], serum Triglycerides) | Measured on weeks 0, 12, 24, and 48.
  To evaluate any beneficial changes in Metabolic Syndrome that may result from probiotic supplementation.
Change in baseline of levels of pro-inflammatory cytokines Interleukin-17 (IL-17), RANKL and Tumor Necrosis Factor (TNF) | Measured on weeks 0, 12, 24, and 48.
  Serum levels may uncover possible anti-inflammatory effects of probiotics
Change from baseline in gut microflora | Measured on weeks 0, 12, 24, and 48.
  Fecal samples will be evaluated for the persistence of the supplemented probiotics in the gut, and their effect on the microbial gut population.
Change from baseline in dual-energy X-ray Absorptiometry (DXA) scans | Measured on weeks 0 and 48.
  To assess bone health by measuring BMD.
Change from baseline in the Fracture Risk Assessment Tool (FRAX) | Measured on weeks 0 and 48.
  To estimate an individual's fracture risk.
Change from baseline in levels of bone resorption and bone formation markers (serum C-terminal telopeptide [CTx], serum procollagen type I N propeptide [PINP], osteocalcin, and bone-specific alkaline phosphatase [BAP]). | Measured on weeks 0, 12, 24, and 48.
  To assess bone health using blood samples.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Altus Research, Lake Worth, Florida
  - Health Awareness Inc., Port Saint Lucie, Florida
  - NeuroTrials Research Inc., Atlanta, Georgia
  - Viable Research, Henderson, Nevada
  - Albuquerque Clinical Trials, Albuquerque, New Mexico

IPD SHARING:
Plan to Share IPD: No